CLINICAL TRIAL: NCT05095922
Title: Effect of Heart-Protecting Musk Pill on Diabetic Microangiopaemia in Type 2 Diabetes Patients
Brief Title: Effect of HMP on Diabetic Microangiopaemia in T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMP2008007p
Record Dates: First submitted 2021-09-28; First posted 2021-10-27 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Angiopathies
Keywords: Heart-protecting musk pill; type 2 diabetes; diabetic angiopathies
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Angiopathies | interventions — Valsartan; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: The type 2 diabetes subjects with diabetic microangiopathy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart-Protecting Musk Pill group (Experimental): Heart-Protecting Musk Pill (pill, 45mg, three times a day, 3 months)+Valsartan Capsules(capsule, 80mg, once a day, 3 months）+Calcium Dobesilate Capsules (capsule, 500mg, three times a day, 3 months)
  Interventions: Drug: Heart-Protecting Musk Pill; Drug: Valsartan Capsules; Drug: Calcium Dobesilate Capsules
- Control group (Placebo Comparator): Valsartan Capsules(capsule, 80mg, once a day, 3 months), Calcium Dobesilate Capsules (capsule, 500mg, three times a day, 3 months)
  Interventions: Drug: Valsartan Capsules; Drug: Calcium Dobesilate Capsules

INTERVENTIONS:
Drug: Heart-Protecting Musk Pill — Heart-Protecting Musk Pill (pill, 45mg, three times a day, 3 months)
  Other Names: Heart-Protecting Musk Pill，National Medicine Permission Number Z31020068，86900674000453
  Arms: Heart-Protecting Musk Pill group
Drug: Valsartan Capsules — Valsartan Capsules(capsule, 80mg, once a day, 3 months）
  Other Names: Valsartan Capsules，National Medicine Permission Number H20040217，86900100000095
Drug: Calcium Dobesilate Capsules — Calcium Dobesilate Capsules(capsule, 500mg, three times a day, 3 months)
  Other Names: Doxium，H20140641

SUMMARY:
The study mainly investigates the therapeutic effect of Heart-Protecting Musk Pill (HMP) on patients with diabetic microangiopathy. According to the indicators of diabetic nephropathy (DN), diabetic retinopathy (DR), oxidative stress and inflammatory factor in patients with diabetic microvascular disease after using HMP, the investigators aim to evaluate the effect of HMP on diabetic microangiopathy, oxidative stress and inflammation.

DETAILED DESCRIPTION:
Diabetes can lead to many diseases as diabetic macrovascular and microvascular complications which result in high disability and mortality rate, thereby seriously affecting the quality of life and life expectancy of diabetic patients. It not only aggravates the family burden of patients, but also becomes the main burden of public health services around the world.

Diabetic nephropathy (DN) and diabetic retinopathy (DR) are more serious in diabetic microangiopathy. The glomerulus and retina have the similar tissue structure and physiological function. Therefore, when they are exposured to the same risk factors can lead to microcirculation damage of kidney and retina. DN and DR have similar pathogenesis and development processes. Although the susceptibility genes and cytokines of DN and DR are different, the two can still be predictors of each other and they often coexist in diabetic patients.

At present, there are few drugs with definite curative effect on the treatment of diabetic microangiopathy, therefore the treatment of diabetic microangiopathy is an aspect that urgently needs a breakthrough in chronic complications of diabetes. Traditional Chinese medicine has a history of preventing and treating diabetes for thousands of years. For the treatment of chronic complications of diabetes by Chinese medicine, although there are not many Chinese medicines that have obtained curative effects, it has indeed accumulated rich experience in the process of research and clinical treatment that Western medicine could not obtain. Therefore, seeking Chinese medicine to effectively treat diabetic microvascular disease has become a direction worthy of attention and research.

Heart-Protecting Musk Pill (HMP) is a commonly used drug in clinical treatment, which comprises seven medicinal substances: Radix Ginseng, Venenum Bufonis, Styrax, Calculus Bovis Artifactus, Cortex Cinnamomi, Borneolum Syntheticum and Artificial Moschus. HMP is a traditional Chinese medicinal compound, which has been effectively used for treating coronary heart disease (CHD) and diabetic macrovascular disease. However, studies on Chinese medicines that are partially similar to HMP have shown that they can improve diabetic retinopathy. Therefore, the study of the efficacy of HMP on diabetic microangiopathy is extremely valuable. Previous researches have shown that HMP owns the effects of reducing oxidative stress, improving inflammation, anti-plateleting aggregation, promoting plasmin activity, and improving hemodynamics. It is possible that HMP can delay or improve the occurrence and development of diabetic microangiopathy through the above effects and even other unclear mechanisms.

At present, the drugs used for clinical treatment of type 2 diabetic microangiopathy are limited. Although the pharmacological indications of HMP can be used to deal with the pathogenesis of diabetic microvascular complications, there is still no clinical study of HMP for the treatment of diabetic microvascular complications. Therefore, this study compared the differences in indicators related to diabetic nephropathy, diabetic retinopathy, oxidative stress, and inflammatory factors between the control group and the HMP group before and after treatment to clarify the therapeutic effect of HMP on diabetic microangiopaemia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Diabetes mellitus
* Prescribed for Valsartan Capsules and Calcium Dobesilate Capsules

Exclusion Criteria:

* Type 1 diabetes mellitus
* Secondary diabetes
* Malignant tumors
* Active infection
* Acute diabetic complications
* Macrovascular complications
* Mental illness
* Intellectual disability
* Impaired heart function
* Impaired liver function
* Impaired kidney function

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Concentration of biochemical Indicators | Change from Baseline TC, TG, HDL-C, LDL-C, FBG, BUN at 3 months
  Total cholesterol(TC), Triglycerides(TG), High-density lipoprotein cholesterol(HDL-C), Low-density lipoprotein cholesterol(LDL-C), Fasting blood glucose(FBG), Blood urea nitrogen(BUN)
Concentration of Glycosylated hemoglobin | Change from Baseline HbA1c at 3 months
  Glycosylated hemoglobin(HbA1c)
Concentration of hypersensitive-c-reactive-protein and Cystatin C | Change from Baseline hs-CRP and CysC at 3 months
  hypersensitive-c-reactive-protein(hs-CRP), Cystatin C(CysC)
Concentration of Serum creatinine | Change from Baseline Scr at 3 months
  Serum creatinine(Scr)
Rate of estimated Glomerular Filtration | Change from Baseline eGFR at 3 months
  estimated Glomerular Filtration Rate(eGFR)
Ratio of Urinary albumin to creatinine | Change from Baseline UACR at 3 months
  Urinary albumin to creatinine Ratio(UACR)
Concentration of Serum fatty acid binding protein 4 | Change from Baseline FABP4 at 3 months
  Serum fatty acid binding protein 4（FABP4)
Indicators of diabetic retinopathy | Change from Baseline effect at 3 months
  The vision and fundus photography will be checked by an ophthalmologist to determine the effect.
Concentration of inflammation indicator | Change from Baseline TNF-α at 3 months
  Tumor Necrosis Factor-α(TNF-α)
Concentration of inflammation indicator | Change from Baseline VEGF at 3 months
  Vascular Endothelial Growth Factor(VEGF)
Concentration of inflammation indicator | Change from Baseline CCL3 at 3 months
  CC chemokine ligand 3(CCL3)
Concentration of Oxidative stress indicator | Change from Baseline SOD at 3 months
  Superoxide dismutase(SOD)
Concentration of Oxidative stress indicator | Change from Baseline GSH-Px at 3 months
  Glutathione peroxidase(GSH-Px)
Concentration of Oxidative stress indicator | Change from Baseline ROS at 3 months
  Reactive oxygen species(ROS）
Clinical characteristics | Change from Baseline Height, Waistline at 3 months
  Height, Waistline
Clinical characteristic | Change from Baseline Weight at 3 months
  Weight
Blood pressure | Change from Baseline SBP, DBP at 3 months
  Systolic Blood Pressure(SBP), Diastolic Blood Pressure(DBP)

CONTACTS AND LOCATIONS:
Overall Officials: Xinlei Wang, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Saaddine JB, Chou CF, Cotch MF, Cheng YJ, Geiss LS, Gregg EW, Albright AL, Klein BE, Klein R. Prevalence of diabetic retinopathy in the United States, 2005-2008. JAMA. 2010 Aug 11;304(6):649-56. doi: 10.1001/jama.2010.1111. PMID 20699456
- [Background] Geraldes P, King GL. Activation of protein kinase C isoforms and its impact on diabetic complications. Circ Res. 2010 Apr 30;106(8):1319-31. doi: 10.1161/CIRCRESAHA.110.217117. PMID 20431074
- [Background] Deng X, Sun L, Lai X, Xiang L, Li Q, Zhang W, Zhang L, Sun S. Tea Polypeptide Ameliorates Diabetic Nephropathy through RAGE and NF-kappaB Signaling Pathway in Type 2 Diabetes Mice. J Agric Food Chem. 2018 Nov 14;66(45):11957-11967. doi: 10.1021/acs.jafc.8b04819. Epub 2018 Nov 1. PMID 30354109
- [Background] Lu L, Qin Y, Chen C, Zhang X, Xu X, Lv C, Wan X, Ruan W, Guo X. The atheroprotective roles of heart-protecting musk pills against atherosclerosis development in apolipoprotein E-deficient mice. Ann Transl Med. 2019 Dec;7(23):714. doi: 10.21037/atm.2019.12.22. PMID 32042730
- [Background] Fan X, Shi M, Wang Y, Liang Q, Luo G. Transcriptional profiling analysis of HMP-treated rats with experimentally induced myocardial infarction. J Ethnopharmacol. 2011 Sep 1;137(1):199-204. doi: 10.1016/j.jep.2011.05.010. Epub 2011 May 13. PMID 21605651